CLINICAL TRIAL: NCT03852407
Title: Allogeneic Hematopoietic Cell Transplantation From HLA-matched Donor After Flu-Mel-PTCy Versus Flu-Mel-ATG Reduced-intensity Conditioning: a Phase II Randomized Study From the Belgian Hematology Society (BHS)
Brief Title: Allogeneic Hematopoietic Cell Transplantation From HLA-matched Donor After Flu-Mel-PTCy Versus Flu-Mel-ATG Reduced-intensity Conditioning
Acronym: HLA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Belgian Hematological Society (Other)
Responsible Party: Principal Investigator, Frédéric Baron, Professor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BHS-TC14; 2017-000824-91 (EudraCT Number)
Record Dates: First submitted 2019-01-21; First posted 2019-02-25 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Acute Myeloid Leukemia in Remission; Myelodysplastic Syndromes; Chronic Myeloid Leukemia in Remission; Myeloproliferative Syndrome; Myeloproliferative Disorder; Acute Lymphoid Leukemia in Remission; Multiple Myeloma; Chronic Lymphoid Leukemia; Non Hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: hematological malignancies; Graft versus host disease; GVHD; Progression free survival; Allogeneic hematopoeitic cell transplantation; HLA-matched donor; reduced intensity conditioning; Overall survival; ATG PK; Immunosuppressive regimen; Prophylaxis
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Multiple Myeloma; Leukemia, B-Cell; Lymphoma, Non-Hodgkin; Hodgkin Disease; Hematologic Neoplasms; Graft vs Host Disease | interventions — thymoglobulin; Melphalan; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fludarabine-Melphalan-Cyclophosphamide (Experimental): FM-PTCy conditioning will consist in IV fludarabine 30 mg/m2 on days -6, -5, -4, -3, and -2 (total dose 150 mg/m2), melphalan given at the dose of 100 mg/m2 on day -2, and cyclophosphamide 50 mg/kg on days +3 and +4.
  Interventions: Drug: Melphalan; Drug: Fludarabine; Drug: Cyclophosphamid
- Fludarabine-Melphalan-thymoglobulin (Experimental): FM-ATG conditioning will consist in IV fludarabine 30 mg/m2 on days -6, -5, -4, -3, and -2 (total dose 150 mg/m2), melphalan given at the dose of 100 mg/m2 on day -2, and ATG (Thymoglobulin®, Genzyme), at a dose of 2.5 mg/kg/d on days -2 and -1.
  Interventions: Drug: Thymoglobulin; Drug: Melphalan; Drug: Fludarabine

INTERVENTIONS:
Drug: Thymoglobulin — ATG: 2.5 mg /kg/day on day -2 and -1 (day 0 is allogenic transplantation)
  Other Names: ATG
  Arms: Fludarabine-Melphalan-thymoglobulin
Drug: Melphalan — 100mg/m² on day -2
  Other Names: alkeran
Drug: Fludarabine — 30mg/m² on days -6, -5, -4, -3, and -2
Drug: Cyclophosphamid — 50 mg/kg on days +3 and +4.
  Other Names: PTCy
  Arms: Fludarabine-Melphalan-Cyclophosphamide

SUMMARY:
The present project aims at comparing two conditioning regimens (FM-PTCy vs FM-ATG). The hypothesis is that one or the two regimens will lead to a 2-year cGRFS rate improvement from 30% (the cGRFS rate with FM without ATG/PTCy) to 45% (Pick-a-winner phase 2 randomized study).

DETAILED DESCRIPTION:
This study is a multicenter, randomized, open-label, phase II study pick-a-winner study, comparing 2 conditioning regimens. A total of 114 eligible patients with HLA-matched donors will be randomized 1:1 between the FM-PTCy arm and the FM-ATG arm, with stratification for donor type (related or unrelated). The recruitment period is 3 years with a 5-year follow-up plus a 10-year additional long-term follow-up (for GVHD status, disease status, second malignancy and QOL). The whole study will be completed within 18 years.

ELIGIBILITY:
Inclusion Criteria:

Patients V.1.1. Diseases

Hematological malignancies confirmed histologically:

* AML in morphological CR or not in morphological CR but not rapidly progressing (i.e. no need to give treatments such as hydroxyurea to maintain WBC count < 10 000 x109/mL);
* MDS;
* CML in CP or AP;
* MPD not in blast crisis,
* MDS/MPD overlap,
* ALL in CR;
* Multiple myeloma;
* CLL;
* Non-Hodgkin's lymphoma (aggressive NHL should have chemosensitive disease);
* Hodgkin's disease with chemosensitive disease or responding to checkpoint inhibitors.

  * Clinical situations

  • Theoretical indication for a standard allo-transplant, but not feasible because:
* Age > 50 yrs;
* Unacceptable end organ performance;
* The physician's decision;
* The patient's decision

  * Underlying 'lower risk' disease, for which Reduced Intensity Conditioning is preferred (eg CLL, MCL)

    * Other inclusion criteria
  * Male or female; fertile patients must use a reliable contraception method;
  * Age 18-75 yrs (children of any age are not allowed in the protocol);
  * Informed consent given by patient or his/her guardian if indicated.

Donors

* Male or female;
* Any age;
* Human Leukocyte Antigen (HLA)-identical sibling donor or 10 of 10 (HLA-A, -B, -C, -DRB1, and -DQB1) HLA allele matched unrelated donor;
* Weight > 15 Kg (because of leukapheresis);
* Fulfills criteria for allogeneic Peripheral Blood Stem Cell (PBSC) donation according to standard procedures;
* Informed consent given by donor or his/her guardian if indicated, as per donor center standard procedures.

Exclusion Criteria:

Patients

* Any condition not fulfilling inclusion criteria;
* Human Immunodeficiency Virus positive;
* Non-hematological malignancy(ies) (except non-melanoma skin cancer) active < 3 years before Hematopoietic Cell Transplantation (HCT).
* Life expectancy severely limited by disease other than malignancy;
* Central Nervous System involvement with disease refractory to intrathecal chemotherapy.
* Terminal organ failure, except for renal failure (dialysis acceptable)

  1. Cardiac: Symptomatic coronary artery disease; ejection fraction <40%; uncontrolled arrhythmia, uncontrolled hypertension;
  2. Pulmonary: Diffusing Capacity of the Lung for Carbon Monoxide (DLCO)< 40% and/or receiving supplementary continuous oxygen, Forced Expiratory Volume in 1 Second (FEV1)< 40%;
  3. Hepatic: Fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin >3 mg/dL, and symptomatic biliary disease;
* Uncontrolled infection;
* Karnofsky Performance Score <70%;
* Patient is a fertile man or woman who is unwilling to use contraceptive techniques during and for 12 months following treatment;
* Patient is a female who is pregnant or breastfeeding;
* Any condition precluding the use of melphalan or Thymoglobulin;

Donors

* Any condition not fulfilling inclusion criteria;
* Unable to undergo leukapheresis because of poor vein access or other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2033-11-01 (Estimated); Study Completion 2038-11-01 (Estimated)

PRIMARY OUTCOMES:
Current GVHD-free, relapse-free survival (cGRFS) | 15 years (the primary endpoint will be first assessed after 191 events have been reached)
  To assess the current GVHD-free, relapse-free survival (cGRFS) for patients in the 2 arms

SECONDARY OUTCOMES:
cGRFS according donor | 15 years
  To assess cGRFS for patients conditioned with FM-PTCy or FM-ATG separately in those transplanted with a related or an unrelated donor
Relapse/progression rate | 15 years
  To assess the relapse/progression rate for patients conditioned with FM-PTCy or FM-ATG
Rate aGVHD | 6 months
  To assess rate of grade II-IV and III-IV acute GVHD (Graft-versus-host disease) in patients conditioned with FM or FM-ATG.
Rate cGVHD | 24 months
  To assess rate of grade of moderate-severe chronic GVHD in patients conditioned with FM or FM-ATG.
Rate of Nonrelapse Mortality (NRM) | 15 years
  To assess rate of Nonrelapse Mortality in patients conditioned with FM-PTCy or FM-ATG.
Rate of Leukemia Free Survival (LFS) | 15 years
  To assess rate of Leukemia Free Survival in patients conditioned with FM-PTCy or FM-ATG.
Rate of Overall Survival (OS) | 15 years
  To assess rate of Overall Survival in patients conditioned with FM-PTCy or FM-ATG.
Proportion of patients alive | 15 years
  To assess the proportion of patients alive without active disease and without systemic immunosuppression

OTHER OUTCOMES:
Hematopoietic engraftment | 2 years
  To assess hematopoietic (whole blood and T cell chimerism) engraftment in the 2 arms.
Quality of immunologic reconstitution | 5 years
  To assess the quality of immunologic reconstitution in the 2 arms
Timing of immunologic reconstitution | 5 years
  To assess the timing (days) of immunologic reconstitution in the 2 arms
Incidences of bacterial infections | 1 year
  To assess the incidences of bacterial infections (number of episode, site, grade) in the 2 arms, in the whole group of patients
Incidences of fungal infections | 1 year
  To assess the incidences of fungal infections (number of episode, site, grade) in the 2 arms, in the whole group of patients
Incidences of viral infections | 1 year
  To assess the incidences of viral infections (number of episode, site, grade) in the 2 arms, in the whole group of patients
Assess Thymoglobulin (ATG) Pharmacokinetic | 10 days
  To assess kinetics of functional ATG serum levels (mg/L) in the FM-ATG arm
Assess ATG Pharmacokinetic in association with cGRFS | 15 years
  To assess kinetics of functional ATG serum levels (mg/L) in the FM-ATG arm in association with cGRFS
Assess ATG Pharmacokinetic in association with NRM | 15 years
  To assess kinetics of functional ATG serum levels (mg/L) in the FM-ATG arm in association with NRM
Assess ATG Pharmacokinetic in association with OS | 15 years
  To assess kinetics of functional ATG serum levels (mg/L) in the FM-ATG arm in association with OS
Assess ATG Pharmacokinetic in association with Relapse/progression | 15 years
  To assess kinetics of functional ATG serum levels (mg/L) in the FM-ATG arm in association with Relapse/progression
Assess ATG Pharmacokinetic in association with Infections | 1 years
  To assess kinetics of functional ATG serum levels (mg/L) in the FM-ATG arm in association with Infections
Assess ATG Pharmacokinetic in association with immunologic reconstitution | 5 years
  To assess kinetics of functional ATG serum levels (mg/L) in the FM-ATG arm in association with immunologic reconstitution (CD4 and NAIVE T cells counts)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Baron, MD,Ph, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (10):
- Belgium (10):
  - ZNA Stuivenberg, Antwerp
  - AZ Sint Jan Brugge, Bruges
  - IJ Bordet, Brussels
  - UZ Brussel, Brussels
  - UCL St Luc, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
  - AZ Delta Roeselare, Roeselare
  - CHU UCL Namur Godinne, Yvoir